CLINICAL TRIAL: NCT05689450
Title: Probability of Optimal Target Attainment of Amikacin in Patients With Febrile Neutropenia During Treatment for a Hematological Disorder: a Prospective, Single-centre Study and PKPD-analysis
Brief Title: Probability of Optimal Target Attainment of Amikacin in Patients With Febrile Neutropenia During Treatment for a Hematological Disorder
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-01218; am23Osthoff
Record Dates: First submitted 2023-01-04; First posted 2023-01-19 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Febrile Neutropenia (FN)
Keywords: Amikacin; Hematological disorder; Aminoglycoside (AG); Area under the curve (AUC); Acute kidney injury (AKI); Pharmacokinetics and pharmacodynamics (PKPD) analysis; Peak serum concentration (Cmax); Trough serum concentration (Cmin); Renal toxicity; Pharmacological target attainment; Amikacin concentration
MeSH Terms: conditions — Febrile Neutropenia; Hematologic Diseases; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection: Amikacin concentration — Blood samples for the measurement of the concentration and calculation of the AUC of amikacin are collected 60 min (+/-30 min) and 8 h (+/-1 h) after the beginning of amikacin infusion. The blood collection after the start of the amikacin infusion will be repeated during every subsequent amikacin administration, but max. during 3 consecutive days.

SUMMARY:
The present trial is a single center, prospective, observational pharmacokinetics and pharmacodynamics (PKPD) cohort study investigating whether patients suffering from a hematological disorder and treated with amikacin due to febrile neutropenia (FN) achieve the predefined amikacin target concentration (Cmax ≥60 mg/L).

DETAILED DESCRIPTION:
Amikacin is an aminoglycoside (AG) that exerts a rapid bactericidal effect against many Gram-negative pathogens. Its pharmacological effect depends on the peak concentration achieved. However, a common side effect of AG is dose-dependent acute kidney injury (AKI), especially when administered over several days due to an accumulation of the drug in the proximal renal tubular cells. In patients in advanced stage of a hematological disease, low body weight influences amikacin pharmacokinetics and pharmacodynamics (PKPD) and increases its clearance. However, there is little known about amikacin PKPD in patients with febrile neutropenia (FN). Whereas the therapeutic efficacy is associated with the peak concentration of AG, toxicity of AG depends on the area under the curve (AUC) or trough level of the drug. When using the AUC to predict renal toxicity, an AUC between 200 and 300 mg/L * h of amikacin has been proposed as a potential threshold for renal toxicity. At the University Hospital Basel (USB), amikacin is administered intravenously (iv) as once daily infusion combined with cefepime or piperacillin/tazobactam immediately after the occurrence of a fever spike in patients with FN. After the iv administration of amikacin, peak concentration is achieved after 30-60 min. The in-house guidelines recommend the administration of lower amikacin dosages compared to other published studies (15 mg/kg body weight vs. 20 mg/kg or up to 30 mg/kg). It remains unclear if adequate peak concentrations are achieved in patients with FN, when lower amikacin doses are administered. The aim of this study is to investigate the probability of optimal pharmacological target attainment (Cmax ≥60 mg/L) during amikacin treatment among patients with FN treated for hematological disorder in order to evaluate the in-house amikacin dosage recommendations. The current project includes the sampling of biological material during hospital admission and the collection of health-related personal data.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Informed consent (IC) as documented by signature
* Documented hematological disorder
* Hospitalization at the USB due to the treatment for a hematological disorder (e.g. chemotherapy, stem cell transplantation)
* Being at risk of developing FN during the hospital stay (e.g. because of chemotherapy)

Exclusion Criteria:

* Previous enrolment into the current study
* Outpatients
* Patients undergoing hemodialysis
* Women who are pregnant (special pharmacokinetic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients being at risk of developing FN after treatment for a hematological disorder, admitted to the Department of Internal Medicine or the Department of Hematology at the University Hospital Basel (USB) and who are intended to receive amikacin iv during their hospital stay will be screened for eligibility.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Change in pharmacological target attainment (Cmax ≥60 mg/L) in blood during amikacin treatment | 60 minutes (+/-30 minutes) and 8 hours (+/-1 hour) after the beginning of amikacin infusion on day 1, day 2 and day 3
  Percentage of patients with optimal pharmacological target attainment (Cmax ≥60 mg/L) in blood during amikacin treatment

SECONDARY OUTCOMES:
AUC >200 mg/L and AUC >300 mg/L* h during amikacin treatment | Up to 3 days after the beginning of amikacin infusion
  Percentage of patients achieving the threshold of potential renal toxicity defined as AUC >200 mg/L and AUC >300 mg/L* h respectively during amikacin treatment
Percentage of patients achieving a calculated Cmin <4 mg/L in blood | Up to 3 days after the beginning of amikacin infusion
  Percentage of patients achieving a calculated Cmin <4 mg/L in blood during amikacin treatment
Incidence of Acute kidney injury (AKI) | Within 7 days after application of amikacin
  Incidence of AKI
Percentage of patients with optimal pharmacological target attainment | Up to 3 days after the beginning of amikacin infusion
  Percentage of patients with optimal pharmacological target attainment using a Cmax/minimal inhibitory concentration (MIC) ≥8 in patients with an identified causative pathogen
Time interval between the detection of the first fever spike and the administration of amikacin | One time assessment at baseline (Day 1)
  Time interval between the detection of the first fever spike and the administration of amikacin

CONTACTS AND LOCATIONS:
Overall Officials: Michael Osthoff, PD Dr. med., Principal Investigator — University Hospital Basel, Division of Internal Medicine
Locations (1):
- University Hospital Basel, Division of Internal Medicine, Basel, Switzerland